CLINICAL TRIAL: NCT06672445
Title: A Phase 1 Placebo-Controlled Dose Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ARO-ATXN2 in Adult Subjects With Spinocerebellar Ataxia Type 2
Brief Title: Study of ARO-ATXN2 Injection in Adults With Spinocerebellar Ataxia Type 2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROATXN2-1001; UTN U111-1308 5875 (Other: WHO); 2024-514763-25 (EudraCT Number)
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Spinocerebellar Ataxia Type 2
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-ATXN2 (Experimental): ARO-ATXN2 Injection
  Interventions: Drug: ARO-ATXN2 Injection
- Placebo (Placebo Comparator): (0.9% NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-ATXN2 Injection — single dose of ARO-ATXN2 by intrathecal (IT) administration
  Arms: ARO-ATXN2
Drug: Placebo — calculated volume to match active treatment by IT administration
  Arms: Placebo

SUMMARY:
Adult participants with spinocerebellar ataxia type 2 (SCA2) who carry ≥33 cytosine, adenine, guanine (CAG) repeats in the ATXN2 gene, and who have met all protocol eligibility criteria will be randomized to receive a single dose of ARO-ATXN2 or placebo and be evaluated for safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating
* Diagnosis of symptomatic SCA2 and ≥33 CAG repeats in the ATXN2 gene based on source verifiable medical records or genetic testing at Screening
* Scale of Assessment and Rating of Ataxia (SARA) score ≤14
* Subjects of childbearing potential must agree to use highly effective contraception in addition to a condom during the study and for at least 90 days following the end of the study or last dose of study drug, whichever is later. Subjects must not donate sperm or eggs during the study and for at least 90 days following the end of the study or last dose of study drug whichever is later

Exclusion Criteria:

* Uncontrolled hypertension (blood pressure >160/100 mmHg)
* History of having received stem cell therapy
* Clinically significant cardiac, liver, or renal disease
* Human immunodeficiency virus (HIV) infection (seropositive at Screening)
* Seropositive for hepatitis B (HBV) or hepatitis C (HCV) at Screening
* Intellectual disability or significant behavioral neuropsychiatric manifestation
* Any contraindications to lumbar puncture, including INR >1.4, platelet count <100,000, and use of anticoagulant or antiplatelet medications that cannot be safely interrupted
* Presence of an implanted shunt for drainage of CSF or an implanted central nervous system (CNS) catheter

Note: Additional inclusion/exclusion criteria may apply per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment -Emergent Adverse Events (TEAEs) Over Time | Through End of Study (EOS), Day 253

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-ATXN2: Maximum Observed Plasma Concentration (Cmax) | Through 24 hours post-dose
PK of ARO-ATXN2: Time to Maximum Observed Plasma Concentration (Tmax) | Through 24 hours post-dose
PK of ARO-ATXN2: Area Under the Plasma Concentration Versus Time Curve from Zero to 24 Hours (AUC0-24) | Through 24 hours post-dose
PK of ARO-ATXN2: Area Under the Plasma Concentration Versus Time Curve from Zero to the Last Quatifiable Plasma Concentration (AUClast) | Through 24 hours post-dose
PK of ARO-ATXN2: Area Under the Plasma Concentration Versus Time Curve from Zero to Infinity (AUCinf) | Through 24 hours post-dose
PK of ARO-ATXN2: Elimination Half-life (t1/2) | Through 24 hours post-dose
PK of ARO-ATXN2: Apparent Systemic Clearance (CL/F) | Through 24 hours post-dose
PK of ARO-ATXN2: Recovery of Unchanged Drug Excreted in Urine (Ae) | Through 24 hours post-dose
PK of ARO-ATXN2: Renal Clearance (CLr) | Through 24 hours post-dose
Percentage of Administered Drug Recovered in Urine | Through 24 hours post-dose
Change from Baseline in Total Protein in Cerebral Spinal Fluid (CSF) Over Time | Baseline through End of Study (EOS), Day 253
Change from Baseline in Glucose in CSF Over Time | Baseline through End of Study (EOS), Day 253
Change from Baseline in Cell Count in CSF Over Time | Baseline through End of Study (EOS), Day 253

CONTACTS AND LOCATIONS:
Locations (16):
- Australia (2):
  - Research Site 8, Sydney, New South Wales
  - Research Site 7, Melbourne, Victoria
- Canada (3):
  - Research Site 2, Montreal, Quebec
  - Research Site 1, Montreal, Quebec
  - Research Site 9, Edmonton
- Research Site 15, Paris, Paris, France
- Germany (2):
  - Research Site 13, Tübingen, Baden-Wurttemberg
  - Research Site 14, Ulm, Baden-Wurttemberg
- Research Site 16, Milan, Italy
- New Zealand (2):
  - Research Site 4, Auckland
  - Research Site 3, Christchurch
- Spain (3):
  - Research Site 10, Barcelona
  - Research Site 11, Barcelona
  - Research Site 12, Seville
- Taiwan (2):
  - Research Site 5, Kaohsiung City
  - Research Site 6, Taipei

IPD SHARING:
Plan to Share IPD: No